CLINICAL TRIAL: NCT01707420
Title: Preoperative Gabapentin for Reduction of Post-tonsillectomy Pain in Children
Brief Title: Preoperative Gabapentin for Post-tonsillectomy Pain in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11-1687
Record Dates: First submitted 2012-10-12; First posted 2012-10-16 (Estimated); Results first posted 2021-01-15 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2020-12

CONDITIONS: Post Operative Pain Management in Children With Tonsillectomy/Adenoidectomy
Keywords: pediatric pain; post operative pain; opioids; emergence agitation; preoperative anxiety; pharmacogenomics
MeSH Terms: conditions — Pain, Postoperative; Emergence Delirium | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gabapentin (Active Comparator): gabapentin, 20 mg/kg, single dose, 60 min prior to surgery
  Interventions: Drug: Gabapentin
- liquid placebo (Placebo Comparator): subjects randomized to the liquid placebo arm will receive a single dose elixir of 0.4 mL/kg given 60 min prior to surgery
  Interventions: Drug: liquid placebo

INTERVENTIONS:
Drug: Gabapentin — The active comparator, Gabapentin, is a structural analog of g-aminobutyric acid which has anticonvulsant properties. This study is a prospective randomized double-blinded trial examining the effectiveness of a single dose of liquid Gabapentin given 60 minutes prior to surgery for pain management in pediatric tonsillectomy/adenoidectomy pediatric patients.
  Other Names: Neurontin
  Arms: Gabapentin
Drug: liquid placebo — Subjects randomized to the liquid placebo will receive an identical appearing liquid placebo of 0.4mL/kg.
  Arms: liquid placebo

SUMMARY:
The typical post-operative course for children following surgical removal of their tonsils and adenoids can be challenging, especially for pain control. First line medications for pain include intravenous and enteral narcotics, acetaminophen and nonsteroidal anti-inflammatory drugs (NSAIDs) or N-methyl-D-aspartate (NMDA) antagonists but their effects appear to be short-lived. Gabapentin has been shown in adult studies to tone down the body's response to pain and decreases opioid use post-operatively. The purpose of this study is to see if a single preoperative dose will reduce post-operative pain scores and the amount of analgesic used.

DETAILED DESCRIPTION:
This is a randomized, double blind, placebo-controlled trial to study the effect of a preoperative oral dose of gabapentin on postoperative analgesic requirements and subjective pain levels in children undergoing tonsillectomy with adenoidectomy. Investigators will also look for a limited set of genotypic variations to explain any difference between individuals or groups in their response to the medication. Additionally, investigators will document potential adverse effects including excessive sedation, respiratory issues, surgical bleeding and emergence agitation/delirium.

Investigators hypothesize that gabapentin will reduce opioid analgesic requirements and pain scores up to 36 hours post adenotonsillectomy without increased adverse effects such as emergence delirium, respiratory complications or bleeding. The clinical effect may depend on the individual's pharmacogenetic profile to look for a specific set of genetic polymorphisms that relate to the metabolism and effect of the study drug, gabapentin, and opioid analgesic pain medications.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for outpatient tonsillectomy and adenoidectomy
* < 60 Kg, between 5th and 95th percentile for weight
* ability to self-report pain
* complete pain diary with assistance from parent or guardian

Exclusion Criteria:

* require pre-anesthesia medication for anxiety
* require interpreter for verbal or written communication
* Obstructive sleep apnea significant enough to not qualify for outpatient surgery per surgeon
* ongoing oxygen dependence, pulmonary hypertension
* elevated risk of regurgitation
* history of seizures
* currently taking psychoactive medications or having a psychiatric condition requiring medications
* chronic pain disorders requiring medications
* renal disease
* developmental or cognitive disabilities
* history of adverse reactions to components of liquid gabapentin or placebo

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2012-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Notides, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Group: Participants received placebo prior to tonsillectomy
- Gabapentin Group: Participants received gabapentin prior to tonsillectomy
Period: Overall Study
Arm/Group | Placebo Group | Gabapentin Group
Started | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo group
- Gabapentin: Gabapentin
- Total: Total of all reporting groups
Arm/Group | Placebo | Gabapentin | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Customized [Median (Full Range); unit: years]
  Median age (years) | 8.0 [5 to 14] | 8.0 [5 to 15] | 8.0 [5 to 15]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 26
  Male | 6 | 4 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 17 | 18 | 35
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: Total Oral Analgesia Consumption
Description: Total mean oral analgesic requirement (cumulative hydrocodone dose (mg/kg)) at nine time points between 0 and 36 hrs post operatively.
Time Frame: Up to 36 hours
Population: Healthy children aged 5 - 16 years old.
Measure: Mean (Standard Deviation); unit: cumulative hydrocodone (mg/kg)
Arm/Group | Placebo Group | Gabapentin Group
Number analyzed (Participants) | 18 | 18
cumulative hydrocodone (mg/kg)
  cumulative hydrocodone (mg/kg) at 36h | 0.228 (0.106) | 0.224 (0.165)
  cumulative hydrocodone (mg/kg) at 24h | 0.200 (0.107) | 0.193 (0.148)
  cumulative hydrocodone (mg/kg) at 12h | 0.171 (0.079) | 0.165 (0.116)
  cumulative hydrocodone (mg/kg) at 8h | 0.157 (0.067) | 0.132 (0.086)
  cumulative hydrocodone (mg/kg) at 4h | 0.135 (0.060) | 0.109 (0.066)
  cumulative hydrocodone (mg/kg) at 1.5h | 0.127 (0.060) | 0.087 (0.066)
  cumulative hydrocodone (mg/kg) at 1h | 0.121 (0.067) | 0.087 (0.066)
  cumulative hydrocodone (mg/kg) at 0.5h | 0.107 (0.077) | 0.068 (0.046)
  cumulative hydrocodone (mg/kg) at 0h | 0.079 (0.077) | 0.011 (0.033)

2. Secondary Outcome: Self-report Pain Score at Rest
Description: Self-report pain scores at rest, using Bieri Faces Scale-Revised. The Bieri Faces Scale-Revised is a patient-reported measure in which patients indicate their pain level by selecting a face with an expression corresponding to their level of pain. Scores range from 0 to 10, with higher scores indicating worse pain. Pain was assessed at eight time points ranging from 0.5 to 36 hours post op.
Time Frame: Up to 36 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Gabapentin Group: The gabapentin (treatment) group was given gabapentin, at a single dose of 20 mg/kg, 60 min prior to surgery in liquid form of less than 0.4 mL/kg total volume.
  This study is a prospective randomized double-blinded trial examining the effectiveness of a single dose of liquid gabapentin given 60 minutes prior to surgery for post-op pain management in healthy pediatric tonsillectomy/adenoidectomy patients.
- Placebo Group: Participants randomized to the placebo arm will received a single dose of placebo, an identical appearing mixture of sweetener, thickener, and water of equal volume, also given 60 min prior to surgery.
Arm/Group | Gabapentin Group | Placebo Group
Number analyzed (Participants) | 18 | 18
score on a scale
  0.5 hours | 5.33 (2.94) | 5.08 (2.71)
  1.0 hours | 4.33 (2.74) | 5.80 (4.02)
  1.5 hours | 4.00 (2.45) | 3.60 (3.30)
  4 hours | 3.46 (2.70) | 3.00 (2.28)
  8 hours | 3.91 (2.57) | 2.71 (1.93)
  12 hours | 2.69 (2.34) | 4.20 (2.35)
  24 hours | 3.04 (2.32) | 4.61 (2.96)
  36 hours | 1.95 (1.74) | 4.00 (1.07)

3. Secondary Outcome: Self-report Pain Score When Swallowing
Description: Self-report pain scores when swallowing using Bieri Faces Scale-Revised. The Bieri Faces Scale-Revised is a patient-reported measure in which patients indicate their pain level by selecting a face with an expression corresponding to their level of pain. Scores range from 0 to 10, with higher scores indicating worse pain. Pain was assessed at eight time points ranging from 0 to 36 hours post op.
Time Frame: Up to 36 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Gabapentin Group | Placebo Group
Number analyzed (Participants) | 18 | 18
score on a scale
  0.5 Hours | 6.47 (3.16) | 5.42 (3.37)
  1 Hours | 4.78 (2.95) | 6.00 (3.65)
  1.5 Hours | 5.40 (3.71) | 5.50 (2.99)
  4 Hours | 4.30 (1.64) | 4.27 (3.44)
  8 Hours | 5.30 (2.67) | 4.00 (2.18)
  12 Hours | 3.86 (2.27) | 4.80 (2.86)
  24 Hours | 5.46 (2.88) | 5.65 (3.64)
  36 Hours | 3.70 (2.41) | 5.13 (2.47)

ADVERSE EVENTS:
Groups:
- Gabapentin: Gabapentin group
Arm/Group | Placebo | Gabapentin
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 3/18 | 9/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=18) | Gabapentin (N=18)
Unplanned admission post tonsillectomy (Surgical and medical procedures) | 1 (1) | 7 (7) — Participants were scheduled for outpatient, same-day surgery. We tracked the number of patients from each group that needed to be admitted, unplanned, to the inpatient hospital unit post-op for any reason.
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No